CLINICAL TRIAL: NCT01511770
Title: Comparative,Randomized,Single-dose,2-way Crossover Bioavailability Study of Dr.Reddy's Laboratories Limited Fluconazole Tablets 200 mg and PFIZER (DIFLUCAN) 200 MG in Healthy Males Under Fasting Condition.
Brief Title: Bioavailability Study of Fluconazole Tablets 200 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA01660
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Fluconazole; Crossover
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluconazole (Experimental): Fluconazole Tablets 200 mg of Dr. Reddy's Laboratories limited.
  Interventions: Drug: Fluconazole
- Diflucan (Active Comparator): Diflucan 200 mg fluconazole tablets of Pfizer
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Fluconazole Tablets, 200 mg
  Other Names: Dr. Reddy's Laboratories
  Arms: Fluconazole
Drug: Fluconazole — Fluconazole 200 mg tablets
  Other Names: Diflucan (Pfizer)
  Arms: Diflucan

SUMMARY:
The objective of this study was an open-label, randomized, 2-way crossover to compare the single-dose relative bioavailability of Dr. Reddy's Laboratories, Ltd. and Pfizer (Diflucan®) 200 mg fluconazole tablets under fasting conditions.

DETAILED DESCRIPTION:
Detailed Description : The study was conducted as an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 18 healthy adult male volunteers. A total of 17 subjects completed the clinical phase of the study. In each period, subjects were housed from the morning dosing until after the 72-hour blood draw. Single oral 200 mg doses were separated by a washout period of 21 days.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

History or presence of significant:

• cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.

In addition, history or presence of:

* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to fluconazole or other azoles. Subjects who have used any drugs or other substances known to be strong inhibitors of CYP (cytochrome P450) enzymes within 10 days prior to first dose.

Subjects who have used any drugs or other substances known to be strong inducers of CYP (cytochrome P450) enzymes within 28 days prior to first dose.

Subjects who have been on an abnormal diet (for whatever reason) during the 28 days prior to the first dosing.

Subjects who, through completion of the study, would have donated in excess of:

* 500 mL of blood in 14 days, or
* 500 - 750 mL of blood in 14 days (unless approved by the Principal Investigator),
* 1000 mL of blood in 90 days,
* 1250 mL of blood in 120 days,
* 1500 mL of blood in 180 days,
* 2000 mL of blood in 270 days,
* 2500 mL of blood in 1 year. Subjects who have participated in another clinical trial within 28 days prior to the first dosing.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2002-08; Primary Completion 2002-08 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | pre dose, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 3.5,4, 6, 9, 12, 24, 48 and 72 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Cohen Street, Saint-laurent, Montreal (quebec), Canada